CLINICAL TRIAL: NCT03167255
Title: A Phase II, Open-Label, Extension Study to Assess the Safety and Efficacy of NS-065/NCNP-01 in Boys With Duchenne Muscular Dystrophy (DMD)
Brief Title: Extension Study of NS-065/NCNP-01 in Boys With Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NS Pharma, Inc. (Industry)
Collaborators: Nippon Shinyaku Co., Ltd. (Industry); Cooperative International Neuromuscular Research Group (Network); Therapeutic Research in Neuromuscular Disorders Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NS-065/NCNP-01-202
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Low Dose cohort of 40 mg/kg and High Dose cohort of 80 mg/kg
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NS-065/NCNP-01 40mg/kg (Experimental): Patients receiving 40mg/kg in the NS-065-NCNP-201 study will continue their current dose for an additional 192 weeks or until enrollment in a separate long-term follow up program of NS-065/NCNP-01, whichever is earlier.
  Interventions: Drug: NS-065/NCNP-01
- NS-065/NCNP-01 80mg/kg (Experimental): Patients receiving 80mg/kg in the NS-065-NCNP-201 study will continue their current dose for an additional 192 weeks or until enrollment in a separate long-term follow up program of NS-065/NCNP-01, whichever is earlier.
  Interventions: Drug: NS-065/NCNP-01

INTERVENTIONS:
Drug: NS-065/NCNP-01 — Received during weekly intravenous infusions

SUMMARY:
This is an open-label, extension study of NS-065/NCNP-01 administered intravenously once weekly for an additional 192 weeks to boys with DMD who complete Study NS-065/NCNP-01-201.

DETAILED DESCRIPTION:
This is a Phase II, multicenter, open-label, extension study of NS-065/NCNP-01 administered intravenously once weekly for an additional 192 weeks to boys with DMD who complete Study NS-065/NCNP-01-201. This study will evaluate the safety, tolerability, and clinical efficacy of NS-065/NCNP-01 at dose levels of up to 80 mg/kg/week administered by weekly IV infusion over an additional treatment period of 192 weeks or until enrollment in a separate long-term follow up program of NS-065/NCNP-01, whichever is earlier.

Patients who complete the Phase II Dose-finding Study NS-065/NCNP-01-201 are eligible to enroll.

ELIGIBILITY:
Inclusion Criteria:

1. Completed Study NS-065/NCNP-01-201 through Week 25.
2. Willing and able to comply with scheduled visits, investigational product administration plan, and study procedures.
3. Stable dose of glucocorticoid (GC), and is expected to remain on the stable dose for the duration of the study.

Exclusion Criteria:

1. Serious or severe adverse event in Study NS-065/NCNP-01-201 that precludes safe use of NS-065/NCNP-01.
2. Patient had a treatment which was made for the purpose of dystrophin or its related protein induction after completion of Study NS-065/NCNP-01-201.
3. Patient took any other investigational drugs after completion of Study NS-065/NCNP-01-201.
4. Patient was judged by the investigator and/or the Sponsor that it was not appropriate to participate in the extension study for other reasons.

Ages: 4 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula R. Clemens, MD, Study Chair — University of Pittsburgh
Locations (6):
- United States (5):
  - UC Davis, Sacramento, California
  - Lurie Children's Hospital, Chicago, Illinois
  - Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 6 sites in the United States and Canada from July 6, 2017 and August 25, 2018.
Pre-assignment Details: Participants who completed study: NS-065/NCNP-01-201 (NCT02740972) were eligible to enroll in this long-term extension study.
Groups:
- NS-065/NCNP-01 40mg/kg: Patients who received 40mg/kg in the NS-065-NCNP-201 study, continued the same treatment with 40mg/kg once weekly for 192 weeks in this extension study.
  NS-065/NCNP-01: Received during weekly intravenous infusions
- NS-065/NCNP-01 80mg/kg: Patients who received 80mg/kg in the NS-065-NCNP-201 study, continued the same treatment with 80mg/kg once weekly for 192 weeks in this extension study.
  NS-065/NCNP-01: Received during weekly intravenous infusions
Period: Overall Study
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population included all participants who received at least one dose of NS-065/NCNP-01 Injection 250 mg infusion in both the Study 201 and extension study (NS-065/NCNP-01-202)
Groups:
- NS-065/NCNP-01 40mg/kg: NS-065/NCNP-01 40mg/kg dose once a week for up to 192 weeks.
  Baseline of Study NS-065/NCNP-01-202: Defined as the measurement taken on Study NS-065/NCNP-01-201 Week 25.
- NS-065/NCNP-01 80mg/kg: NS-065/NCNP-01 80mg/kg dose once a week for up to 192 weeks.
  Baseline of Study NS-065/NCNP-01-202: Defined as the measurement taken on Study NS-065/NCNP-01-201 Week 25.
- Total: Total of all reporting groups
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.0 (1.75) | 7.8 (2.11) | 7.9 (1.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 25.0 (4.95) | 23.0 (6.72) | 24.0 (5.79)
Height [Mean (Standard Deviation); unit: cm] | 115.9 (7.54) | 115.3 (9.96) | 115.6 (8.54)
Body Mass Index(BMI) [Mean (Standard Deviation); unit: kg/m^2] | 18.4 (2.17) | 17.0 (2.54) | 17.7 (2.39)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Time to Stand (TTSTAND) Versus Matched Historical Controls
Description: A primary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): Time to Stand (TTSTAND)
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157, 205 in Study 202
Population: The analysis population included all participants who received at least one dose of investigational drug. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: seconds
Groups:
- NS-065/NCNP-01 40mg/kg: NS-065/NCNP-01 40mg/kg dose once a week for up to 192 weeks.
  Baseline of Study NS-065/NCNP-01-202: Defined as the measurement taken on Study NS-065/NCNP-01-201 Week 25 Visit.
- NS-065/NCNP-01 80mg/kg: NS-065/NCNP-01 80mg/kg dose once a week for up to 192 weeks.
  Baseline of Study NS-065/NCNP-01-202: Defined as the measurement taken on Study NS-065/NCNP-01-201 Week 25 Visit.
- Total NS-065/NCNP-01 Group: All 16 patients who received treatment with NS-065/NCNP-01 were included in the Full Analysis Set population.
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
seconds
  Week 37 | 0.17 (1.60) | -0.38 (1.59) | -0.11 (1.12)
  Week 49: number analyzed (Participants) | 8 | 7 | 15
  Week 49 | 0.69 (1.60) | -0.60 (1.61) | 0.07 (1.13)
  Week 73: number analyzed (Participants) | 7 | 7 | 14
  Week 73 | 0.55 (1.63) | 0.03 (1.62) | 0.29 (1.14)
  Week 109: number analyzed (Participants) | 7 | 7 | 14
  Week 109 | 0.77 (1.68) | 0.30 (1.67) | 0.54 (1.18)
  Week 157: number analyzed (Participants) | 5 | 6 | 11
  Week 157 | 1.32 (1.80) | 1.45 (1.72) | 1.44 (1.23)
  Week 205: number analyzed (Participants) | 6 | 7 | 13
  Week 205 | 1.62 (1.82) | 3.58 (1.70) | 2.71 (1.24)

2. Primary Outcome: Change From Baseline in Time to Stand (TTSTAND) Velocity Versus Matched Historical Controls
Description: A primary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): Time to Stand (TTSTAND) Velocity
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157, 205 in Study 202
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: rise/s
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
rise/s
  Week 37 | 0.03 (0.03) | 0.04 (0.03) | 0.04 (0.02)
  Week 49: number analyzed (Participants) | 8 | 7 | 15
  Week 49 | 0.03 (0.03) | 0.04 (0.03) | 0.04 (0.02)
  Week 73: number analyzed (Participants) | 7 | 7 | 14
  Week 73 | 0.03 (0.03) | 0.50 (0.03) | 0.04 (0.02)
  Week 109: number analyzed (Participants) | 7 | 7 | 14
  Week 109 | 0.04 (0.03) | 0.04 (0.03) | 0.04 (0.02)
  Week 157: number analyzed (Participants) | 5 | 6 | 11
  Week 157 | 0.02 (0.04) | -0.05 (0.03) | -0.01 (0.02)
  Week 205: number analyzed (Participants) | 7 | 7 | 14
  Week 205 | -0.02 (0.03) | -0.07 (0.03) | -0.04 (0.02)

3. Primary Outcome: Number of Participants With Treatment Related Adverse Events as Assessed by CTCAE v4.0.
Description: For adverse events (AEs) starting in study 201 (NCT02740972) which are not resolved at the time of enrollment into this study 202, any change in outcome or relatedness were reported in study 201.
  For AEs starting in study 201 which increase in severity or becomes serious after enrollment in this study 202, a new AE was reported in this study.
  Treatment-emergent AEs (TEAEs) were summarized by dose level. Coding was done by system organ class and preferred term (using the Medical Dictionary for Regulatory Activities (MedDRA)). Level of severity was assessed using the CTCAE grading system.
Time Frame: Up to 192 weeks of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
Participants
  Participants with TEAE | 8 | 8 | 16
  Participants with drug-related TEAE | 0 | 1 | 1
  Participants with CTCAE ≥ Grade 3 | 0 | 2 | 2
  Participants with TEAEs leading to discontinuation | 0 | 0 | 0
  Participants with serious TEAE | 1 | 2 | 3
  Death | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Time to Run/Walk 10 Meters Test (TTRW) Versus Matched Historical Controls
Description: A secondary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): Time to Run/Walk 10 meters test (TTRW)
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157, 205 in Study 202
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
seconds
  Week 37 | -0.41 (1.06) | -1.35 (1.05) | -0.88 (0.75)
  Week 49: number analyzed (Participants) | 8 | 7 | 15
  Week 49 | -0.87 (1.06) | -0.74 (1.06) | -0.82 (0.75)
  Week 73 | -1.15 (1.06) | -0.68 (1.05) | -0.91 (0.75)
  Week 109 | -0.67 (1.06) | -0.25 (1.05) | -0.46 (0.75)
  Week 157: number analyzed (Participants) | 7 | 7 | 14
  Week 157 | 0.13 (1.07) | 0.56 (1.06) | 0.35 (0.75)
  Week 205: number analyzed (Participants) | 6 | 8 | 14
  Week 205 | 0.89 (1.10) | 2.84 (1.05) | 2.00 (0.76)

5. Secondary Outcome: Change From Baseline in Time to Run/Walk 10 Meters Test (TTRW) Velocity Versus Matched Historical Controls
Description: A secondary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): Time to Run/Walk 10 meters test (TTRW) Velocity.
  The results were converted into velocity (meter/time).
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157, 205 in Study 202
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
m/s
  Week 37 | 0.15 (0.17) | 0.53 (0.17) | 0.34 (0.12)
  Week 49: number analyzed (Participants) | 8 | 7 | 15
  Week 49 | 0.35 (0.17) | 0.28 (0.17) | 0.32 (0.12)
  Week 73 | 0.44 (0.17) | 0.28 (0.17) | 0.36 (0.12)
  Week 109 | 0.33 (0.17) | 0.12 (0.17) | 0.23 (0.12)
  Week 157: number analyzed (Participants) | 7 | 7 | 14
  Week 157 | 0.24 (0.18) | -0.02 (0.17) | 0.11 (0.12)
  Week 205: number analyzed (Participants) | 6 | 8 | 14
  Week 205 | 0.14 (0.18) | -0.23 (0.17) | -0.06 (0.13)

6. Secondary Outcome: Change From Baseline in Time to Climb 4 Stairs (TTCLIMB) Versus Matched Historical Controls
Description: A secondary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): Time to Climb 4 stairs (TTCLIMB)
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157, 205 in Study 202
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
seconds
  Week 37 | -0.37 (1.54) | 0.38 (1.54) | 0.01 (1.09)
  Week 49: number analyzed (Participants) | 8 | 6 | 14
  Week 49 | -0.26 (1.54) | 0.28 (1.56) | 0.02 (1.09)
  Week 73 | -0.08 (1.54) | 0.44 (1.54) | 0.18 (1.09)
  Week 109 | 1.02 (1.54) | 1.08 (1.54) | 1.05 (1.09)
  Week 157: number analyzed (Participants) | 7 | 7 | 14
  Week 157 | 4.28 (1.55) | 2.95 (1.55) | 3.61 (1.09)
  Week 205: number analyzed (Participants) | 6 | 7 | 13
  Week 205 | 3.00 (1.66) | 3.18 (1.58) | 3.16 (1.14)

7. Secondary Outcome: Change From Baseline in Time to Climb 4 Stairs (TTCLIMB) Velocity Versus Matched Historical Controls
Description: A secondary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): Time to Climb 4 stairs (TTCLIMB) Velocity. The results were converted into velocity (meter/time).
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157, 205 in Study 202
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
m/s
  Week 37 | 0.04 (0.04) | 0.01 (0.04) | 0.02 (0.03)
  Week 49: number analyzed (Participants) | 8 | 6 | 14
  Week 49 | 0.05 (0.04) | 0.01 (0.04) | 0.03 (0.03)
  Week 73 | 0.06 (0.04) | 0.03 (0.04) | 0.05 (0.03)
  Week 109 | 0.03 (0.04) | -0.02 (0.04) | 0.00 (0.03)
  Week 157: number analyzed (Participants) | 7 | 7 | 14
  Week 157 | 0.04 (0.04) | -0.07 (0.04) | -0.01 (0.03)
  Week 205: number analyzed (Participants) | 6 | 7 | 13
  Week 205 | 0.05 (0.05) | -0.07 (0.04) | -0.01 (0.03)

8. Secondary Outcome: Change From Baseline in North Star Ambulatory Assessment (NSAA) Score Versus Matched Historical Controls
Description: A secondary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): North Star Ambulatory Assessment (NSAA) score
  The NSAA is a functional scale devised for use in ambulant children with Duchenne muscular dystrophy (DMD).
  It consists of 17 activities graded 0 (unable to perform), 1 (performs with modifications), 2 (normal movement). It assesses abilities necessary to remain ambulant that have been found to progressively deteriorate in untreated DMD patients, as well as in other muscular dystrophies such as Becker Muscular Dystrophy. NSAA Total Score ranges from 0 to 34, with a score of 34 implying normal function.
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157 in Study 202
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
score on a scale
  Week 37 | 2.53 (1.83) | -0.02 (1.83) | 1.27 (1.29)
  Week 49: number analyzed (Participants) | 8 | 7 | 15
  Week 49 | 1.91 (1.83) | 0.14 (1.85) | 1.05 (1.29)
  Week 73 | 0.41 (1.83) | 1.23 (1.83) | 0.83 (1.29)
  Week 109 | 0.91 (1.83) | 1.36 (1.83) | 1.14 (1.29)
  Week 157: number analyzed (Participants) | 7 | 7 | 14
  Week 157 | -1.31 (1.85) | 0.35 (1.85) | -0.47 (1.30)

9. Secondary Outcome: Change From Baseline in Six-Minute Walk Test (6MWT) Versus Matched Historical Controls
Description: A secondary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): Six-Minute Walk Test (6MWT)
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157 in Study 202
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: m
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
m
  Week 37: number analyzed (Participants) | 8 | 7 | 15
  Week 37 | 15.15 (26.84) | 13.03 (28.15) | 14.30 (19.29)
  Week 49: number analyzed (Participants) | 8 | 6 | 14
  Week 49 | 9.90 (26.84) | 16.94 (29.70) | 13.32 (19.75)
  Week 73 | -0.73 (26.84) | 18.14 (26.89) | 8.72 (18.87)
  Week 109 | -16.35 (26.84) | 18.51 (26.89) | 1.10 (18.87)
  Week 157: number analyzed (Participants) | 7 | 6 | 13
  Week 157 | -41.61 (28.08) | -27.76 (29.71) | -34.86 (20.28)

10. Secondary Outcome: Change From Baseline in Quantitative Muscle Testing (QMT) for Handgrip Versus Matched Historical Controls
Description: A secondary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): Quantitative Muscle Testing (QMT) for Handgrip For QMT tests, the higher of each of the bilateral scores recorded for each muscle group at each visit were analyzed. QMT tests were analyzed by dominant/non-dominant side.
  QMT is a well-established method for measuring muscle weakness in neuromuscular disease. Patients will be placed on an examination table with a back-support system to eliminate the need for manual back stabilization. Following a single practice administration, each patient will complete a scored QMT evaluation (perform 2 tests; with the higher of the 2 values used for data analysis). QMT will be performed by recording force in pounds through a direct computer interface with a strain gauge.
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157, 205 in Study 202
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: lb
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
lb
  Handgrip, Week 37: number analyzed (Participants) | 8 | 6 | 14
  Handgrip, Week 37 | 0.56 (1.28) | 1.86 (1.42) | 1.09 (0.94)
  Handgrip, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Handgrip, Week 49 | 1.63 (1.28) | 2.34 (1.37) | 1.96 (0.93)
  Handgrip, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Handgrip, Week 73 | 1.85 (1.32) | 0.83 (1.42) | 1.39 (0.96)
  Handgrip, Week 109: number analyzed (Participants) | 8 | 6 | 14
  Handgrip, Week 109 | 2.22 (1.28) | 2.00 (1.42) | 2.12 (0.94)
  Handgrip, Week 157: number analyzed (Participants) | 4 | 4 | 8
  Handgrip, Week 157 | 2.94 (1.55) | 3.10 (1.59) | 3.06 (1.10)
  Handgrip, Week 205: number analyzed (Participants) | 1 | 3 | 4
  Handgrip, Week 205 | 7.34 (2.61) | 4.05 (1.74) | 5.00 (1.39)
  Dominant Side Handgrip, Week 37: number analyzed (Participants) | 8 | 6 | 14
  Dominant Side Handgrip, Week 37 | 0.22 (1.28) | 2.17 (1.42) | 1.03 (0.95)
  Dominant Side Handgrip, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Dominant Side Handgrip, Week 49 | 1.17 (1.28) | 2.70 (1.37) | 1.88 (0.93)
  Dominant Side Handgrip, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Dominant Side Handgrip, Week 73 | 0.99 (1.33) | 1.26 (1.43) | 1.13 (0.96)
  Dominant Side Handgrip, Week 109: number analyzed (Participants) | 8 | 6 | 14
  Dominant Side Handgrip, Week 109 | 1.86 (1.28) | 1.61 (1.43) | 1.76 (0.95)
  Dominant Side Handgrip, Week 157: number analyzed (Participants) | 4 | 4 | 8
  Dominant Side Handgrip, Week 157 | 2.41 (1.57) | 2.66 (1.61) | 2.56 (1.11)
  Dominant Side Handgrip, Week 205: number analyzed (Participants) | 1 | 3 | 4
  Dominant Side Handgrip, Week 205 | 7.37 (2.68) | 4.36 (1.76) | 5.17 (1.42)
  Non-Dominant Side Handgrip, Week 37: number analyzed (Participants) | 8 | 6 | 14
  Non-Dominant Side Handgrip, Week 37 | 1.45 (1.20) | 2.19 (1.32) | 1.79 (0.96)
  Non-Dominant Side Handgrip, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Handgrip, Week 49 | 1.95 (1.20) | 1.99 (1.27) | 1.97 (0.96)
  Non-Dominant Side Handgrip, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Non-Dominant Side Handgrip, Week 73 | 3.38 (1.24) | 0.58 (1.33) | 2.05 (0.98)
  Non-Dominant Side Handgrip, Week 109: number analyzed (Participants) | 8 | 6 | 14
  Non-Dominant Side Handgrip, Week 109 | 3.02 (1.20) | 2.93 (1.33) | 3.08 (0.97)
  Non-Dominant Side Handgrip, Week 157: number analyzed (Participants) | 4 | 4 | 8
  Non-Dominant Side Handgrip, Week 157 | 4.67 (1.47) | 3.01 (1.50) | 3.29 (1.14)
  Non-Dominant Side Handgrip, Week 205: number analyzed (Participants) | 1 | 3 | 4
  Non-Dominant Side Handgrip, Week 205 | 3.92 (2.53) | 4.48 (1.65) | 2.94 (1.38)

11. Secondary Outcome: Change From Baseline in Quantitative Muscle Testing (QMT) for Elbow Flexors Versus Matched Historical Controls
Description: A secondary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): Quantitative Muscle Testing (QMT) for Elbow Flexors For QMT tests, the higher of each of the bilateral scores recorded for each muscle group at each visit were analyzed. QMT tests were analyzed by dominant/non-dominant side.
  QMT is a well-established method for measuring muscle weakness in neuromuscular disease. Patients will be placed on an examination table with a back-support system to eliminate the need for manual back stabilization. Following a single practice administration, each patient will complete a scored QMT evaluation (perform 2 tests; with the higher of the 2 values used for data analysis). QMT will be performed by recording force in pounds through a direct computer interface with a strain gauge.
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157, 205 in Study 202
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: lb
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
lb
  Elbow Flexors, Week 37: number analyzed (Participants) | 8 | 7 | 15
  Elbow Flexors, Week 37 | -0.11 (0.72) | 0.57 (0.78) | 0.21 (0.53)
  Elbow Flexors, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Elbow Flexors, Week 49 | 0.57 (0.72) | 0.63 (0.78) | 0.60 (0.53)
  Elbow Flexors, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Elbow Flexors, Week 73 | -0.70 (0.75) | 0.82 (0.81) | 0.00 (0.55)
  Elbow Flexors, Week 109: number analyzed (Participants) | 8 | 7 | 15
  Elbow Flexors, Week 109 | 0.53 (0.72) | 0.30 (0.78) | 0.42 (0.53)
  Elbow Flexors, Week 157: number analyzed (Participants) | 4 | 5 | 9
  Elbow Flexors, Week 157 | -0.24 (0.89) | 1.05 (0.85) | 0.49 (0.61)
  Elbow Flexors, Week 205: number analyzed (Participants) | 3 | 4 | 7
  Elbow Flexors, Week 205 | 0.74 (0.98) | 0.07 (0.91) | 0.34 (0.66)
  Dominant Side Elbow Flexors, Week 37: number analyzed (Participants) | 8 | 7 | 15
  Dominant Side Elbow Flexors, Week 37 | -0.01 (0.77) | 0.39 (0.83) | 0.18 (0.56)
  Dominant Side Elbow Flexors, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Dominant Side Elbow Flexors, Week 49 | 0.48 (0.77) | -0.38 (0.83) | 0.08 (0.56)
  Dominant Side Elbow Flexors, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Dominant Side Elbow Flexors, Week 73 | -0.53 (0.80) | 0.97 (0.86) | 0.16 (0.58)
  Dominant Side Elbow Flexors, Week 109: number analyzed (Participants) | 8 | 7 | 15
  Dominant Side Elbow Flexors, Week 109 | 0.71 (0.77) | 0.14 (0.83) | 0.44 (0.56)
  Dominant Side Elbow Flexors, Week 157: number analyzed (Participants) | 4 | 5 | 9
  Dominant Side Elbow Flexors, Week 157 | 0.00 (0.94) | 0.31 (0.91) | 0.20 (0.65)
  Dominant Side Elbow Flexors, Week 205: number analyzed (Participants) | 3 | 4 | 7
  Dominant Side Elbow Flexors, Week 205 | 0.77 (1.04) | 0.20 (0.97) | 0.46 (0.70)
  Non-Dominant Side Elbow Flexors, Week 37: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Elbow Flexors, Week 37 | 0.42 (0.68) | 0.84 (0.73) | 0.61 (0.50)
  Non-Dominant Side Elbow Flexors, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Elbow Flexors, Week 49 | 0.44 (0.68) | 1.02 (0.73) | 0.71 (0.50)
  Non-Dominant Side Elbow Flexors, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Non-Dominant Side Elbow Flexors, Week 73 | -0.45 (0.71) | 0.60 (0.76) | 0.02 (0.52)
  Non-Dominant Side Elbow Flexors, Week 109: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Elbow Flexors, Week 109 | 0.65 (0.68) | -0.21 (0.73) | 0.25 (0.50)
  Non-Dominant Side Elbow Flexors, Week 157: number analyzed (Participants) | 4 | 5 | 9
  Non-Dominant Side Elbow Flexors, Week 157 | -0.15 (0.85) | 1.52 (0.81) | 0.80 (0.59)
  Non-Dominant Side Elbow Flexors, Week 205: number analyzed (Participants) | 3 | 4 | 7
  Non-Dominant Side Elbow Flexors, Week 205 | 0.47 (0.95) | -0.45 (0.87) | -0.07 (0.64)

12. Secondary Outcome: Change From Baseline in Quantitative Muscle Testing (QMT) for Elbow Extensors Versus Matched Historical Controls
Description: A secondary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): Quantitative Muscle Testing (QMT) for Elbow Extensors For QMT tests, the higher of each of the bilateral scores recorded for each muscle group at each visit were analyzed. QMT tests were analyzed by dominant/non-dominant side.
  QMT is a well-established method for measuring muscle weakness in neuromuscular disease. Patients will be placed on an examination table with a back-support system to eliminate the need for manual back stabilization. Following a single practice administration, each patient will complete a scored QMT evaluation (perform 2 tests; with the higher of the 2 values used for data analysis). QMT will be performed by recording force in pounds through a direct computer interface with a strain gauge.
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157, 205 in Study 202
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: lb
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
lb
  Elbow Extensors, Week 37: number analyzed (Participants) | 8 | 7 | 15
  Elbow Extensors, Week 37 | 0.55 (0.73) | 0.88 (0.78) | 0.70 (0.53)
  Elbow Extensors, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Elbow Extensors, Week 49 | 0.48 (0.73) | 0.93 (0.78) | 0.68 (0.53)
  Elbow Extensors, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Elbow Extensors, Week 73 | 0.27 (0.76) | 0.96 (0.81) | 0.60 (0.55)
  Elbow Extensors, Week 109: number analyzed (Participants) | 8 | 7 | 15
  Elbow Extensors, Week 109 | 1.23 (0.73) | -0.05 (0.78) | 0.63 (0.53)
  Elbow Extensors, Week 157: number analyzed (Participants) | 4 | 5 | 9
  Elbow Extensors, Week 157 | 1.56 (0.91) | -0.01 (0.86) | 0.70 (0.62)
  Elbow Extensors, Week 205: number analyzed (Participants) | 3 | 4 | 7
  Elbow Extensors, Week 205 | -0.06 (1.01) | 0.07 (0.92) | 0.06 (0.67)
  Dominant Side Elbow Extensors, Week 37: number analyzed (Participants) | 8 | 7 | 15
  Dominant Side Elbow Extensors, Week 37 | 0.68 (0.76) | 1.21 (0.82) | 0.92 (0.55)
  Dominant Side Elbow Extensors, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Dominant Side Elbow Extensors, Week 49 | 0.54 (0.76) | 0.53 (0.82) | 0.53 (0.55)
  Dominant Side Elbow Extensors, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Dominant Side Elbow Extensors, Week 73 | -1.02 (0.79) | 1.08 (0.85) | -0.05 (0.57)
  Dominant Side Elbow Extensors, Week 109: number analyzed (Participants) | 8 | 7 | 15
  Dominant Side Elbow Extensors, Week 109 | 1.04 (0.76) | -0.07 (0.82) | 0.52 (0.55)
  Dominant Side Elbow Extensors, Week 157: number analyzed (Participants) | 4 | 5 | 9
  Dominant Side Elbow Extensors, Week 157 | 0.78 (0.93) | 0.22 (0.89) | 0.43 (0.64)
  Dominant Side Elbow Extensors, Week 205: number analyzed (Participants) | 3 | 4 | 7
  Dominant Side Elbow Extensors, Week 205 | -0.11 (1.02) | 0.54 (0.95) | 0.25 (0.69)
  Non-Dominant Side Elbow Extensors, Week 37: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Elbow Extensors, Week 37 | 0.48 (0.63) | 0.78 (0.67) | 0.61 (0.46)
  Non-Dominant Side Elbow Extensors, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Elbow Extensors, Week 49 | 0.65 (0.63) | 1.19 (0.67) | 0.90 (0.46)
  Non-Dominant Side Elbow Extensors, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Non-Dominant Side Elbow Extensors, Week 73 | 1.18 (0.66) | 0.74 (0.70) | 0.99 (0.48)
  Non-Dominant Side Elbow Extensors, Week 109: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Elbow Extensors, Week 109 | 1.84 (0.63) | -0.22 (0.67) | 0.87 (0.46)
  Non-Dominant Side Elbow Extensors, Week 157: number analyzed (Participants) | 4 | 5 | 9
  Non-Dominant Side Elbow Extensors, Week 157 | 2.27 (0.81) | -0.01 (0.75) | 1.05 (0.55)
  Non-Dominant Side Elbow Extensors, Week 205: number analyzed (Participants) | 3 | 4 | 7
  Non-Dominant Side Elbow Extensors, Week 205 | 0.74 (0.91) | -0.39 (0.81) | 0.17 (0.61)

13. Secondary Outcome: Change From Baseline in Quantitative Muscle Testing (QMT) for Knee Flexors Versus Matched Historical Controls
Description: A secondary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): Quantitative Muscle Testing (QMT) for Knee Flexors For QMT tests, the higher of each of the bilateral scores recorded for each muscle group at each visit were analyzed. QMT tests were analyzed by dominant/non-dominant side.
  QMT is a well-established method for measuring muscle weakness in neuromuscular disease. Patients will be placed on an examination table with a back-support system to eliminate the need for manual back stabilization. Following a single practice administration, each patient will complete a scored QMT evaluation (perform 2 tests; with the higher of the 2 values used for data analysis). QMT will be performed by recording force in pounds through a direct computer interface with a strain gauge.
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157, 205 in Study 202
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: lb
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
lb
  Knee Flexors, Week 37: number analyzed (Participants) | 8 | 7 | 15
  Knee Flexors, Week 37 | -0.35 (1.48) | 2.04 (1.56) | 0.82 (1.10)
  Knee Flexors, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Knee Flexors, Week 49 | 0.77 (1.48) | 1.20 (1.56) | 1.03 (1.10)
  Knee Flexors, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Knee Flexors, Week 73 | 1.04 (1.50) | 2.33 (1.60) | 1.64 (1.12)
  Knee Flexors, Week 109: number analyzed (Participants) | 8 | 7 | 15
  Knee Flexors, Week 109 | 2.04 (1.48) | 2.73 (1.56) | 2.42 (1.10)
  Knee Flexors, Week 157: number analyzed (Participants) | 4 | 5 | 9
  Knee Flexors, Week 157 | 2.43 (1.70) | 2.68 (1.66) | 3.02 (1.26)
  Knee Flexors, Week 205: number analyzed (Participants) | 3 | 4 | 7
  Knee Flexors, Week 205 | 2.21 (2.09) | 2.87 (1.70) | 2.24 (1.30)
  Dominant Side Knee Flexors, Week 37: number analyzed (Participants) | 8 | 7 | 15
  Dominant Side Knee Flexors, Week 37 | -0.69 (1.46) | 2.06 (1.54) | 0.60 (1.07)
  Dominant Side Knee Flexors, Week 49: number analyzed (Participants) | 8 | 6 | 14
  Dominant Side Knee Flexors, Week 49 | 0.06 (1.46) | 1.77 (1.60) | 0.84 (1.09)
  Dominant Side Knee Flexors, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Dominant Side Knee Flexors, Week 73 | -0.23 (1.51) | 1.99 (1.60) | 0.80 (1.11)
  Dominant Side Knee Flexors, Week 109: number analyzed (Participants) | 8 | 7 | 15
  Dominant Side Knee Flexors, Week 109 | 1.87 (1.46) | 2.63 (1.54) | 2.24 (1.07)
  Dominant Side Knee Flexors, Week 157: number analyzed (Participants) | 4 | 5 | 9
  Dominant Side Knee Flexors, Week 157 | 3.00 (1.76) | 2.26 (1.68) | 2.51 (1.22)
  Dominant Side Knee Flexors, Week 205: number analyzed (Participants) | 3 | 4 | 7
  Dominant Side Knee Flexors, Week 205 | 2.34 (1.93) | 2.78 (1.79) | 2.47 (1.31)
  Non-Dominant Side Knee Flexors, Week 37: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Knee Flexors, Week 37 | -0.78 (1.25) | 2.40 (1.33) | 0.67 (0.92)
  Non-Dominant Side Knee Flexors, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Knee Flexors, Week 49 | 1.04 (1.25) | 1.05 (1.33) | 1.02 (0.92)
  Non-Dominant Side Knee Flexors, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Non-Dominant Side Knee Flexors, Week 73 | 0.93 (1.28) | 1.81 (1.37) | 1.26 (0.95)
  Non-Dominant Side Knee Flexors, Week 109: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Knee Flexors, Week 109 | 1.71 (1.25) | 2.17 (1.33) | 1.90 (0.92)
  Non-Dominant Side Knee Flexors, Week 157: number analyzed (Participants) | 4 | 5 | 9
  Non-Dominant Side Knee Flexors, Week 157 | 1.35 (1.50) | 2.29 (1.44) | 2.20 (1.09)
  Non-Dominant Side Knee Flexors, Week 205: number analyzed (Participants) | 3 | 4 | 7
  Non-Dominant Side Knee Flexors, Week 205 | 2.40 (1.84) | 2.22 (1.49) | 1.86 (1.14)

14. Secondary Outcome: Change From Baseline in Quantitative Muscle Testing (QMT) for Knee Extensors Versus Matched Historical Controls
Description: A secondary efficacy endpoint was compared to Baseline of Study 201 (NCT02740972): Quantitative Muscle Testing (QMT) for Knee Extensors For QMT tests, the higher of each of the bilateral scores recorded for each muscle group at each visit were analyzed. QMT tests were analyzed by dominant/non-dominant side.
  QMT is a well-established method for measuring muscle weakness in neuromuscular disease. Patients will be placed on an examination table with a back-support system to eliminate the need for manual back stabilization. Following a single practice administration, each patient will complete a scored QMT evaluation (perform 2 tests; with the higher of the 2 values used for data analysis). QMT will be performed by recording force in pounds through a direct computer interface with a strain gauge.
Time Frame: Baseline 201, Weeks 37, 49, 73, 109, 157, 205 in Study 202
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: lb
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
lb
  Knee Extensors, Week 37: number analyzed (Participants) | 8 | 7 | 15
  Knee Extensors, Week 37 | 1.25 (1.93) | 1.10 (1.97) | 1.15 (1.38)
  Knee Extensors, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Knee Extensors, Week 49 | 0.04 (1.93) | 1.11 (1.96) | 0.52 (1.37)
  Knee Extensors, Week 73: number analyzed (Participants) | 7 | 7 | 14
  Knee Extensors, Week 73 | -1.00 (1.96) | 2.57 (1.95) | 0.87 (1.38)
  Knee Extensors, Week 109 | 0.89 (1.93) | 1.14 (1.92) | 1.03 (1.36)
  Knee Extensors, Week 157: number analyzed (Participants) | 4 | 6 | 10
  Knee Extensors, Week 157 | 3.01 (2.21) | 0.88 (2.02) | 1.76 (1.55)
  Knee Extensors, Week 205: number analyzed (Participants) | 3 | 4 | 7
  Knee Extensors, Week 205 | 1.16 (2.71) | -0.59 (2.15) | -0.11 (1.62)
  Dominant Side Knee Extensors, Week 37: number analyzed (Participants) | 8 | 7 | 15
  Dominant Side Knee Extensors, Week 37 | -0.81 (1.82) | 1.87 (1.86) | 0.44 (1.30)
  Dominant Side Knee Extensors, Week 49: number analyzed (Participants) | 8 | 6 | 14
  Dominant Side Knee Extensors, Week 49 | 0.33 (1.82) | 2.14 (1.88) | 1.16 (1.30)
  Dominant Side Knee Extensors, Week 73: number analyzed (Participants) | 7 | 7 | 14
  Dominant Side Knee Extensors, Week 73 | -1.45 (1.85) | 1.11 (1.85) | -0.07 (1.30)
  Dominant Side Knee Extensors, Week 109 | 1.19 (1.82) | 0.73 (1.81) | 0.99 (1.28)
  Dominant Side Knee Extensors, Week 157: number analyzed (Participants) | 4 | 6 | 10
  Dominant Side Knee Extensors, Week 157 | 1.00 (2.10) | 1.28 (1.91) | 1.51 (1.47)
  Dominant Side Knee Extensors, Week 205: number analyzed (Participants) | 3 | 4 | 7
  Dominant Side Knee Extensors, Week 205 | 0.63 (2.59) | 1.35 (2.04) | 0.45 (1.55)
  Non-Dominant Side Knee Extensors, Week 37: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Knee Extensors, Week 37 | 1.72 (1.73) | -0.12 (1.86) | 0.86 (1.23)
  Non-Dominant Side Knee Extensors, Week 49: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Knee Extensors, Week 49 | 0.46 (1.73) | 0.20 (1.86) | 0.34 (1.23)
  Non-Dominant Side Knee Extensors, Week 73: number analyzed (Participants) | 7 | 6 | 13
  Non-Dominant Side Knee Extensors, Week 73 | -0.51 (1.78) | 1.03 (1.91) | 0.18 (1.27)
  Non-Dominant Side Knee Extensors, Week 109: number analyzed (Participants) | 8 | 7 | 15
  Non-Dominant Side Knee Extensors, Week 109 | -0.39 (1.73) | 1.99 (1.86) | 0.72 (1.23)
  Non-Dominant Side Knee Extensors, Week 157: number analyzed (Participants) | 4 | 5 | 9
  Non-Dominant Side Knee Extensors, Week 157 | 2.97 (2.10) | 0.42 (2.01) | 1.23 (1.46)
  Non-Dominant Side Knee Extensors, Week 205: number analyzed (Participants) | 3 | 4 | 7
  Non-Dominant Side Knee Extensors, Week 205 | 0.82 (2.57) | -1.67 (2.08) | -0.58 (1.53)

ADVERSE EVENTS:
Time Frame: Up to 192 weeks
Description: Incidence of Adverse Events as assessed by CTCAE v4.0
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/8 | 3/16
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NS-065/NCNP-01 40mg/kg (N=8) | NS-065/NCNP-01 80mg/kg (N=8) | Total NS-065/NCNP-01 Group (N=16)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NS-065/NCNP-01 40mg/kg (N=8) | NS-065/NCNP-01 80mg/kg (N=8) | Total NS-065/NCNP-01 Group (N=16)
Nasopharyngitis (Infections and infestations) | 4 (10) | 5 (16) | 9 (26)
Influenza (Infections and infestations) | 3 (5) | 1 (2) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (5) | 2 (5)
Body tinea (Infections and infestations) | 2 (3) | 0 (0) | 2 (3)
Ear infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Coxsackie viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (9) | 1 (1) | 5 (10)
Arthropod bite (Injury, poisoning and procedural complications) | 4 (5) | 2 (2) | 6 (7)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Incision site swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Incision site vesicles (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Traumatic tooth displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (9) | 10 (16)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 2 (2) | 5 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (3)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (7) | 3 (7) | 6 (14)
Constipation (Gastrointestinal disorders) | 2 (4) | 1 (1) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (4) | 3 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Tooth development disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (21) | 2 (6) | 5 (27)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (6) | 4 (6) | 6 (12)
Catheter site erythema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Catheter site swelling (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Infusion site pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site extravasation (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 1 (1)
Tenderness (General disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Spinal deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 6 (7)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Flat affect (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Body height decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Hypercalciuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The most restrictive relevant agreement on the PI provides that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is not less than 30 days from the time submitted to the sponsor for review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT03167255/Prot_SAP_000.pdf